CLINICAL TRIAL: NCT01489319
Title: Evaluation of the Ovarian Dynamic Response and the Inflammatory Response to Oral Lipid Challenge in Relation to Body Composition in Polycystic Ovary Syndrome
Brief Title: Evaluation of Oral Lipid Ingestion in Relation to Ovarian Androgen Secretion in Polycystic Ovary Syndrome (PCOS)
Acronym: ELI-ROAS
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The PI left Indiana University. The findings served as preliminary data for a recently awarded NIH R01 grant.
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Frank Gonzalez, Associate Professor, Director, Division of Reproductive Endocrinology and Infertility, Indiana University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IU-PCOS-0112
Record Dates: First submitted 2011-12-06; First posted 2011-12-09 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Polycystic Ovary Syndrome
Keywords: inflammation; body composition; hyperandrogenism; insulin resistance
MeSH Terms: conditions — Polycystic Ovary Syndrome; Inflammation; Hyperandrogenism; Insulin Resistance | interventions — salicylsalicylic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (6):
- Nl Wt PCOS - Nl Abdominal Adiposity (Experimental): 10 normal weight women with PCOS who have normal abdominal adiposity established by DEXA
  Interventions: Drug: Salsalate
- Nl Wt PCOS - Increased Abdominal Adiposity (Experimental): 10 normal weight women with PCOS who have increased abdominal adiposity established by DEXA
  Interventions: Drug: Salsalate
- Obese PCOS (No Intervention): 10 obese women with PCOS
- Nl Wt Controls - Nl Abdominal Adiposity (No Intervention): 10 normal weight ovulatory women serving as controls who have normal abdominal adiposity established by DEXA
- Nl Wt Controls - Increased Abdominal Adiposity (No Intervention): 10 normal weight ovulatory women serving as controls who have increased abdominal adiposity established by DEXA
- Obese Controls (No Intervention): 10 obese ovulatory women serving as controls

INTERVENTIONS:
Drug: Salsalate — 4 out of 10 subjects will receive salsalate 2.0 gm twice a day for 12 weeks; 4 out of 10 subjects will receive PCE 200 mg containing 20% resveratrol twice a day for 12 weeks.
  Arms: Nl Wt PCOS - Nl Abdominal Adiposity
Drug: Salsalate — 4 out of the 10 subjects will receive salsalate 2.0 gm twice a day for 12 weeks; 4 out of 10 subjects will receive PCE 200 mg containing 20% resveratrol twice a day for 12 weeks.
  Arms: Nl Wt PCOS - Increased Abdominal Adiposity

SUMMARY:
The purpose of this study is to determine the relationship between lipid-induced inflammation and ovarian androgen secretion in women with polycystic ovary syndrome (PCOS); and to examine the effect of salsalate and polygonum cuspidatum extract (PCE) containing resveratrol on lipid-induced inflammation, ovarian androgen secretion, body composition and ovulation in a subset of normal weight women with PCOS.

DETAILED DESCRIPTION:
The investigator hypothesizes that in women with PCOS, HCG administration will stimulate an exaggerated ovarian androgen response, dairy cream ingestion will stimulate white blood cells to generate an inflammatory response, and that there is a relationship between HCG-stimulated ovarian androgen secretion and the inflammatory response to dairy cream ingestion regardless of body fat status. Thirty (30) women with PCOS (10 normal weight with normal abdominal adiposity, 10 normal weight with increased abdominal adiposity and 10 obese) and 30 ovulatory control women (10 normal weight with normal abdominal adiposity, 10 normal weight with increased abdominal adiposity and 10 obese) will participate over a 3-year period.

The investigator also hypothesizes that both salsalate and PCE administration for 12 weeks will attenuate the ovarian androgen response to HCG administration and the inflammatory response to dairy cream ingestion, reduce abdominal adiposity, increase insulin sensitivity and induce ovulation in normal weight women with PCOS. A subset of 16 women with PCOS of which 8 will receive salsalate (4 normal weight with normal abdominal adiposity and 4 normal weight with increased abdominal adiposity) and 8 will receive PCE (4 normal weight with normal abdominal adiposity and 4 normal weight with increased abdominal adiposity) will participate in this intervention over a 3-year period. This pilot project will help determine the feasibility of conducting a larger double-blind, randomized trial in women with PCOS to further test the latter hypothesis.

ELIGIBILITY:
General Inclusion Criteria:

* Acceptable health based on interview, medical history, physical examination, and lab tests
* Ability to comply with the requirements of the study
* Ability and willingness to provide signed, witnessed informed consent

Inclusion Criteria for PCOS:

* Between the ages of 18-40 years
* Body mass index between 18 and 25, or between 30 and 40
* Less than or equal to 8 periods annually
* An elevated serum androgen level or skin manifestations of androgen excess
* Normal thyroid function tests and normal prolactin level
* Exclusion of late-onset adrenal hyperplasia

Inclusion Criteria for Ovulatory Controls:

* Between the ages of 18-40 years
* Body mass index between 18 and 25, or between 30 and 40
* Normal regular monthly periods
* No clinical evidence of androgen excess
* No evidence of polycystic ovaries on ultrasound

Exclusion Criteria:

* Diabetes mellitus
* Clinically significant pulmonary, cardiac ,renal, hepatic, neurologic, psychiatric, infectious, and malignant disease
* High blood pressure
* Current or recent (within 6 weeks prior to study entry) injection of any drugs known or suspected to affect reproductive function including oral contraceptives, metformin, thiazolidinediones, glucocorticoids, GnRH-agonists, or anti-androgens (spironolactone, flutamide, etc)
* Documented or suspected history of use of recent (within one year) illicit drug abuse or alcoholism
* Tobacco smoking if salsalate or PCE will be administered
* Ingestion of any investigational drugs within 4 weeks prior to study onset
* Pregnancy or lactation (less than or equal to 6 weeks postpartum)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2012-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
White blood cell nuclear factor kappa B (NFkappaB) activation in response to oral lipid ingestion and ovarian androgen secretion in response to human chorionic gonadotropin (HCG) stimulation. | 3 years
  This outcome along with insulin sensitivity derived from an oral glucose tolerance test (OGTT) and body composition measured by dual energy absorptiometry (DEXA) will be assessed in all study subjects (PCOS and controls).

SECONDARY OUTCOMES:
White blood cell NFkappaB activation following oral lipid ingestion in response to 12 weeks of salsalate or PCE administration. | 3 years
  This outcome will be assessed in a subset of normal weight women with PCOS who have either normal (n=4) or increased (n=4) abdominal adiposity.
Ovarian androgen secretion following HCG administration in response to 12 weeks of salsalate or PCE administration. | 3 years
  This outcome will be assessed in a subset of normal weight women with PCOS who have either normal (n=4) or increased (n=4) abdominal adiposity.
Body composition status measured by DEXA in response to 12 weeks of salsalate or PCE administration. | 3 years
  This outcome will be assessed in a subset of normal weight women with PCOS who have either normal (n=4) or increased (n=4) abdominal adiposity.
Insulin sensitivity derived from an OGTT in response to 12 weeks of salsalate or PCE administration. | 3 years
  This outcome will be assessed in a subset of normal weight women with PCOS who have either normal (n=4) or increased (n=4) abdominal adiposity.
Ovulation rates documented by serum progesterone in response to 12 weeks of salsalate or PCE administration | 3 years
  This outcome will be assessed in a subset of normal weight women with PCOS who have either normal (n=4) or increased (n=4) abdominal adiposity.

CONTACTS AND LOCATIONS:
Overall Officials: Frank González, M.D., Principal Investigator — Indiana University
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Gonzalez F, Considine RV, Abdelhadi OA, Acton AJ. Lipid-induced mononuclear cell cytokine secretion in the development of metabolic aberration and androgen excess in polycystic ovary syndrome. Hum Reprod. 2020 May 1;35(5):1168-1177. doi: 10.1093/humrep/deaa056. PMID 32325487
- [Derived] Gonzalez F, Considine RV, Abdelhadi OA, Acton AJ. Inflammation Triggered by Saturated Fat Ingestion Is Linked to Insulin Resistance and Hyperandrogenism in Polycystic Ovary Syndrome. J Clin Endocrinol Metab. 2020 Jun 1;105(6):e2152-67. doi: 10.1210/clinem/dgaa108. PMID 32140727
- [Derived] Gonzalez F, Considine RV, Abdelhadi OA, Acton AJ. Saturated Fat Ingestion Promotes Lipopolysaccharide-Mediated Inflammation and Insulin Resistance in Polycystic Ovary Syndrome. J Clin Endocrinol Metab. 2019 Mar 1;104(3):934-946. doi: 10.1210/jc.2018-01143. PMID 30590569